CLINICAL TRIAL: NCT01127334
Title: Validation of a Robust Method for Kinematic Analysis of Ventricular Mechanical Dyssynchrony by Two Dimensional Echocardiography in Patients With Cardiac Resynchronization Devices for Chronic Systolic Heart Failure and Conduction System Disease
Brief Title: Pilot Study Using Echocardiography to Evaluate Patients With Heart Failure and Dyssynchrony Who Have a CRT-D Device
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator terminated study
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Donny R. Stokes M.D., University of Mississippi Medical Center
Other Study IDs: 2010-0069
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2010-05

CONDITIONS: Systolic Heart Failure
Keywords: Dyssynchrony; Cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Systolic Heart Failure, Dyssynchrony, CRT-D: Patients with systolic heart failure and dyssynchrony that have a CRT-D that have not been optimized in the past 3 months.

SUMMARY:
Out of all the patients that receive a CRT-D ( a dual chamber pacemaker with defibrillator ) for cardiac resynchronization therapy there is approximately one-third that do not respond. We believe that by using a simple technique that includes routine echocardiography that are normally performed in these patients could help us better understand how to program their device to reach better optimization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-110 years
2. Must have a CRT-D (A biventricular pacemaker with defibrillator)
3. Last optimization of their device (CRT-D) must not have been done in the past 3 months
4. Must be optimal heart failure medical regimen. This includes target dose of beta-blocker and angiotensin converting enzyme inhibitor (ACE-I) (or equivalent; i.e angiotensin receptor blocker (ARB); or balanced preload and afterload reducers with hydralazine and nitrates.)

Exclusion Criteria:

1. Less than 18 years of age or greater than 110 years old.
2. Does not have a CRT-D
3. Optimization of their device has occurred in the past 3 months
4. Not on optimal medical therapy for heart failure as listed in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology and electrophysiology clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donny R. Stokes, M.D., Principal Investigator — University of Mississippi Medical Center; John P. Payne, M.D., Study Director — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States